CLINICAL TRIAL: NCT01223482
Title: An Investigation of Women's Experiences Following Karyotyping Products of Conception After a Miscarriage
Brief Title: A Study Looking at Women's Experiences After a Miscarriage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: California State University, Stanislaus (Other)
Collaborators: Stanford University (Other)
Responsible Party: Janey Youngblom, CSU Stanislaus
Other Study IDs: 1011-017
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-09

CONDITIONS: Miscarriage
Keywords: Miscarriage; Karyotyping; Genetic testing
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Miscarriage with genetic testing: This is a study population of women that have had a miscarriage and had genetic testing performed. The investigators would like to know what their experiences were following their miscarriage and testing.
- Miscarriage without genetic testing: This cohort is considered the control group. These women have not had genetic testing done, but are asked questions regarding their miscarriage experience.

SUMMARY:
Studies have shown that a majority of pregnancies that end in miscarriage are due to a chromosome abnormality usually involving a duplicated or missing chromosome. Often this happens by chance and is not likely to occur in future pregnancies. For many women, a miscarriage can be a traumatic experience and can cause feelings of loss and grief. The option of genetic testing, such as karyotyping, may offer an explanation for the miscarriage and may help some women find closure in their loss. However, no literature exists on a women's experience with genetic testing following a miscarriage. This assumption that the knowledge that can be gained from karyotyping may be a positive experience for a woman following a miscarriage should be studied and the results published. This study will address whether routine karyotyping should be offered following a miscarriage for the purpose of benefiting the patient's experience.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for this project will be females, 18 years or older, of any ethnicity that have had a 1st trimester miscarriage within the last one year, who currently reside in the US and have done so for the past one year.

Exclusion Criteria:

* Exclusion criteria will be males, females younger than 18 years of age, females with a miscarriage over one year, non-US residents and US residents where the miscarriage occurred outside of the US.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators are targeting woman based on the inclusion and exclusion criteria provided below.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-02 (Estimated); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Http://Www.Surveymonkey.Com/S/Miscarriagestudy3, Palo Alto, California, United States